CLINICAL TRIAL: NCT05824845
Title: QIST Collaborative - Arthroplasty Research Cohort (ARC) Study - a Collaborative, Longitudinal Observational Cohort Study of Patients Undergoing Primary Hip and Knee Replacements in the United Kingdom
Brief Title: QIST Collaborative - Arthroplasty Research Cohort (ARC) Study
Status: Recruiting | Type: Observational
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: University of York (Other)
Responsible Party: Sponsor
Other Study IDs: ARC Study
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hip Arthritis; Knee Arthritis
Keywords: Hip Replacement; Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ARC Study Cohort
  Interventions: Procedure: Hip/Knee Replacement

INTERVENTIONS:
Procedure: Hip/Knee Replacement — Hip/Knee Replacement

SUMMARY:
The ARC Study is a national observational cohort study to investigate patient reported and clinical outcomes after hip and knee replacements. The study has the following objectives:

1. To evaluate outcomes following hip and knee replacements.
2. To determine risk factors for adverse outcomes in primary hip and knee replacements.
3. To identify targets for future research and intervention in patients undergoing primary hip and knee replacements
4. To provide a resource from which to identify potential participants for future clinical trials, and to use data collected in the ARC Study as comparison or control data for trial participants who have been randomised to receive one or more interventions.

Participants are recruited and consented online. Patients are invited to participate by collaborating surgical teams nationally in outpatient clinics at the time of being added to a waiting list, in addition to an advertising campaign to recruit patients. They are directed to an online portal where they will be able to review further information.

Consent and data collection is completed electronically through patients entering data online. Baseline demographics and characteristics are recorded, including details of socio-demographics, lifestyle, health status and patient reported outcome measures (PROMs). Patients then undergo hip/knee replacement and postoperative rehabilitation according to the standard care and protocols of the hospital and the preferences of their treating surgeon.

Follow-up data, including PROMs, is collected via online questionnaires up to two years following surgery. The study will ultimately also enable multiple trials to be embedded within the cohort study, using a 'Trials within Cohorts' (TwiCs) methodology.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria:

1. UK Resident
2. Able to read and understand documentation and questionnaires in English language
3. Undergoing elective primary hip or knee arthroplasty (THR, TKR or UKR)
4. Age 18 years or over
5. Provides the necessary consents relating to data collection and use of study data, data linkage, future research and invitation to involvement in future trials

Exclusion Criteria:

Provided a participant meets all of the inclusion criteria, there are no exclusion criteria for the cohort study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK Residents age 18 years or over undergoing elective primary hip or knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L health-related quality of life score | 2 years

SECONDARY OUTCOMES:
PROMIS-10 | 2 years
  Patient-Reported Outcomes Measurement Information System Global Health
Oxford Hip Score | 2 years
Oxford Knee Score | 2 years
Musculoskeletal Health Questionnaire | 2 years
  MSK-HQ
Hospital for Special Surgery Hip/Knee Replacement Expectations Surveys | 2 years
  Perception of success/fulfilment of expectations
Patient Health Questionnaire-4 | 2 years
  PHQ-4
11-point Numerical Pain Rating Scale | 2 years
  Pain
Pain Catastrophising Scale | 2 years
Length of stay | 2 years
  Self-reported by study specific electronic questionnaire
Activity | 2 years
  Levels of exercise and activity self-reported by study specific electronic questionnaire
Return to work | 2 years
  Work status self-reported by electronic questionnaire using National Statistics Socio-economic Classification
Readmission within 30 days | 30 days
Surgical Site Infection | 2 years
Periprosthetic Fracture | 2 years
Dislocation | 2 years
Revision/Re-operation | 2 years
Mortality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria Healthcare NHS Foundation Trust, Ashington, United Kingdom

IPD SHARING:
Plan to Share IPD: No